CLINICAL TRIAL: NCT06539702
Title: To Reveal the Predictive Value of Preoperative Hemogram Parameters and BRAF Molecular Test in Predicting Malignancy in Cases With Thyroid Nodules Detected by Bethesda 3 Cytology.
Brief Title: Preoperative Hemogram Parameters and BRAF Molecular Test Detected by Bethesda 3 Cytology.
Acronym: Bethesda3
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: E-48670771-514.99-237222286
Record Dates: First submitted 2024-07-09; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Blood Platelet Disorder; BRAF V600E; Thyroid Nodule; Cytologic Atypia
Keywords: Thyroid; carcinoma; Bethesda 3; BRAF
MeSH Terms: conditions — Blood Platelet Disorders; Thyroid Nodule; Thyroid Diseases; Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Pathological specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2/Group B (Benign), Group M (Malign): Mean Platelet Volume (MPV), Neutrophil/lymphocyte Ratio (NLR), Platelet/Lymphocyte Ratio (PLR) and Lymphocyte/Monocyte Ratio (LMR) will be recorded in preoperative hemograms. Among the patients included in the study, BRAF molecular testing will be performed on the preoperative cytology of 25 patients whose thyroidectomy materials were reported to be malignant. with thyroid nodule identified by Bethesda 3 cytology were examined retrospectively. According to the pathology results, they were divided into 2 groups: benign and malignant.
  Group B (Benign);Preoperative hemogram parameters, Bethesda 3 cytology, Thyroidectomy, benign pathology.
  Group M (Malign);Preoperative hemogram parameters, Betheda 3 cytology, Thyroidectomy, malign pathology, BRAF molecular test

SUMMARY:
The main hypothesis of this study is that preoperative hemogram parameters can be used as biomarkers for malignancy in patients with thyroid nodule Bethesda 3 cytology.

The secondary hypothesis is that BRAF molecular testing has a high predictive value in predicting malignancy in patients with thyroid nodule Bethesda 3 cytology.

Primary outcome: Preoperative hemogram parameters. Secondary outcome: BRAF positivity.

DETAILED DESCRIPTION:
The main hypothesis of this study is that preoperative hemogram parameters can be used as biomarkers for malignancy in patients with thyroid nodule Bethesda 3 cytology.

The secondary hypothesis is that BRAF molecular testing has a high predictive value in predicting malignancy in patients with thyroid nodule Bethesda 3 cytology.

Primary outcome: Preoperative hemogram parameters. Secondary outcome: BRAF positivity. This study aims to reduce unnecessary thyroidectomies, thyroidectomy complications and treatment costs due to Bethesda 3 cytology.

The age and gender of all patients to be included in the study will be recorded. Mean Platelet Volume (MPV), Neutrophil/lymphocyte Ratio (NLR), Platelet/Lymphocyte Ratio (PLR) and Lymphocyte/Monocyte Ratio (LMR) will be recorded in preoperative hemograms. Nodule sizes detected by preoperative Bethesda III cytology will be recorded. The sizes of nodules with preoperative AUS cytology after thyroidectomy, determined as a result of pathological examination, will be recorded. Patients with malignant cytology will be divided into papillary thyroid carcinoma (PTC), Follicular Thyroid Carcinoma (FTC), and tumor sizes will be recorded. Among the patients included in the study, BRAF molecular testing will be performed on the preoperative cytology of 25 patients whose thyroidectomy materials were reported to be malignant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 -75
2. Patients who were diagnosed with Bethesda III as a result of preoperative FNAC and decided to undergo thyroidectomy

Exclusion Criteria:

1. Patients over 18 years old and under 75 years old
2. Patients with malignancy detected in another focus with preoperative Bethesda III FNAC
3. Detection of malignancy in another focus other than the nodule with Bethesda III cytological result after thyroidectomy
4. Failure to obtain preoperative hemogram results Patients who do not agree to participate in scientific studies for BRAF testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 -75
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-08-06 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Mean Platelet Volume (MPV) (fL) | 1 week
  Mean Platelet Volume (MPV) (fL) values will be taken and recorded in the preoperative hemogram parameters of all patients.
Neutrophil/lenfosit Ratio (NLR)(103/µL) | 1 week
  Neutrophil/lymphocyte ratio (NLR) will be calculated by taking the Neutrophil (103/µL) and Lymphocyte (103/µL) values in the preoperative hemogram parameters of all patients.
Platelet/Lenfosit Ratio (PLR)(103/µL) | 1 week
  Platelet/lymphocyte ratio (PLR) will be calculated by taking the Platelet (103/µL) and Lymphocyte (103/µL) values in the preoperative hemogram parameters of all patients.
Lenfosit/Monosit Ratio (LMR)(103/µL) | 1 week
  Lymphocyte/Monocyte Ratio (LMR) will be calculated by taking the Lymphocyte (103/µL) and Monocyte (103/µL) values in the preoperative hemogram parameters of all patients.

SECONDARY OUTCOMES:
BRAF molecular test | 1 week
  Pathological molecular test (25 patients)

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Kesici, Assoc.Prof., Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bostan H, Sencar ME, Calapkulu M, Hepsen S, Akhanli P, Duger H, Ucan B, Kizilgul M, Ozturk Unsal I, Ozbek M, Cakal E. The predictive value of hematologic parameters in the risk of thyroid malignancy in cases with atypia/follicular lesion of undetermined significance. Eur Arch Otorhinolaryngol. 2022 Aug;279(8):4077-4084. doi: 10.1007/s00405-021-07248-9. Epub 2022 Jan 10. PMID 35006341
- [Result] Acar S, Ercetin C, Sahbaz NA, Tutal F, Yapalak Y, Cosan F, Erbil Y. Hemodynamic Instability during Thyroidectomy in Graves' Disease. J Invest Surg. 2022 Mar;35(3):627-631. doi: 10.1080/08941939.2021.1914785. Epub 2021 Apr 28. PMID 33908335